CLINICAL TRIAL: NCT01210183
Title: Biological Response of Stage IV Knee Osteoarthritis to Serial 12.5% Dextrose Injections Without Weight Bearing Restriction: A Double Arthroscopic Assessment
Brief Title: Biological Response of Stage IV Knee Osteoarthritis to Serial 12.5% Dextrose
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Rosario (Other)
Responsible Party: Principal Investigator, Gastón Andrés Topol, Principle Investigator, Universidad Nacional de Rosario
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ProvingCartilageGrowth
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Knee Osteoarthritis
Keywords: Dextrose; Cartilage; Regeneration
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dextrose intraarticularly administered — 9 ml of 12.5% dextrose
  Other Names: Glucose

SUMMARY:
Dextrose injection in end-stage knee arthritis will cause growth of cartilage cells in a particular area of complete cartilage loss. Dextrose concentration will be 12.5%. Cartilage status will be monitored by pre and post treatment arthroscopy views with specialized (methylene blue) staining for cartilage.

DETAILED DESCRIPTION:
Historical, compliance, examination,anesthetic injection, radiographic and arthroscopic screening will be completed. One month after arthroscopy completion, the intervention phase will begin.

INTERVENTION

* Injection of 12.5% dextrose at 0, 1 and 2 months.
* Stand up without using only the non-injected leg for 3 days after each injection.
* Avoid running and squatting as feasible.
* Ensure that the injected knee descends stairs first ascends stairs last for 3 days.
* May take Acetaminophen.
* No NSAIDS for 2 days before and 10 days after a treatment. PRN NSAIDs only.
* No glucosamine or chondroitin should be taken.

SECOND ARTHROSCOPY TIMING

* A minimum of 4 months after first arthroscopy, when schedulable.
* After a minimum of 3 monthly injections of dextrose 12.5% .

METHOD OF ARTHROSCOPY

* Only the medial compartment will be entered to minimize trauma.
* Methylene blue will be applied and allowed to remain in knee for 5 minutes prior to flush.
* A standardized method video scan of the medial femoral compartment will be conducted.
* At second arthroscopy, the area of heaviest cartilage growth, if any, in the base of the Out-IV lesion will be biopsied with a Jamshidi needle at a 45 degree angle. (Limited by the optics of single port entry ).
* Biopsy, if taken, will be sent for decortication to enable specimen to be cut, safranin O application to determine proteoglycan production, polarized light to differentiate fibrous from hyaline cartilage, and immunohistologic straining for Type I and Type Ii cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≤ 90 kilos.
* Available for clinic any day.
* Agreeable to keep coming if pain stops.
* More than one phone number.(close relative ok)
* Willing to wait 6 months prior to considering a TKA.
* Good strength in arms to help stand.
* Knee flexion more than 100 degrees.
* 90% reduction of standing, walking and sitting pain 5 minutes after intraarticular injection of 9 ml of 0.25% dextrose.
* XRay repeat with camera at knee height confirms bone on bone status in the medial compartment.

Exclusion Criteria:

* No dementia.
* No radiating back pain.
* No systemic inflammatory conditions.
* No history of knee fracture or infection.
* No cancer history.
* No blood thinners.
* No daily narcotic.
* No walking limitation from another cause.
* Repetitive squatting or stair use on job.
* Inability to use one arm to help come to stand.
* Painful hip ROM or imitative of patient's pain.
* Knee extension lacking more than 15 degrees on each side.
* Any degree of valgus.
* Varus of 20 degree or more.
* A painful Baker's cyst.
* Visible bone shift when walking
* Meniscal tear seen on arthroscopy that could block motion and needs trimming.
* Significant loose bodies seen on arthroscopy.
* Severe synovitis seen on arthroscopy.
* More than 1 outerbridge lesion in the medial compartment of the femur.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quality of cartilage growth | 0 to 3 months
  A Jamshidi needle biopsy will be obtained at 45 degrees in the area of maximum cartilage growth and analyzed for quality/type of cartilage if such growth is seen.
Number of sections of medial condyle with loss, no change or growth of cartilage. | 7.5 month mean
  Arthroscopy of all 9 sections of the medial condyle for each of 6 knees will be viewed by each of 3 arthroscopers who will render their opinion for each section. They will compare sections from 1st and 2nd arthroscopy side by side, and will be asked to indicate loss of cartilage no change or growth of cartilage for each of sections on each of 6 knees.
  Still photos of the biopsy study site wiThe photo of the Out IV lesion will be analyzed in a blinded fashion for a visual or computerized assessment of the percentage of lesion size covered by cartilage buds.

SECONDARY OUTCOMES:
Walking pain | 0 to 3 years
  Subjects will be asked to estimate their walking pain on a 10 point scale over the preceding 2 weeks.
Flexion range of motion | 0 to 3 months
  The total flexion range of motion of the knee will be measured goniometrically.
WOMAC | 7.5 Months
  WOMAC will be administered at time 0 and at time of the 2nd arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Gaston A Topol, M.D., Principal Investigator — Hospital Provincial de Rosario
Locations (1):
- Hospital Provincial de Rosario, Rosario, Santa Fe Province, Argentina

REFERENCES:
- [Derived] Topol GA, Podesta LA, Reeves KD, Giraldo MM, Johnson LL, Grasso R, Jamin A, Clark T, Rabago D. Chondrogenic Effect of Intra-articular Hypertonic-Dextrose (Prolotherapy) in Severe Knee Osteoarthritis. PM R. 2016 Nov;8(11):1072-1082. doi: 10.1016/j.pmrj.2016.03.008. Epub 2016 Apr 4. PMID 27058744